CLINICAL TRIAL: NCT06781203
Title: Determination of Optimal Sleep Treatment Elements (The DOSE Project) - DISA RCT
Brief Title: Determination of Optimal Sleep Treatment Elements (The DOSE Project) - DISA
Acronym: DISA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); Enversion (Unknown)
Responsible Party: Principal Investigator, Prof. Robert (Bobby) Zachariae, DMSc, MSc, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fort.: 2022-0367531, 2099; 148790 (Other Grant/Funding Number: TrygFonden)
Record Dates: First submitted 2024-09-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Insomnia Chronic
Keywords: hvil
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: In addition to investigator masking, we aim to mask the participants as much as possible. Participants in the intervention group will know that they recieve treatment, whereas participants in the care as usual waitlist control group will receive standard sleep hygiene advice, and be informed that they will receive an offer for treatment upon completed data collection. However, neither group will know that there are other groups involved. Care providers (GPs) are not masked, but any potential bias arising from this is expected to be minimal, as they do not deliver the intervention treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care as usual waitlist control (No Intervention): Waitlist control; care as usual coupled with generic sleep hygiene advice. Access to treatment provided after final measurement.
- Digitally delivered CBTI (eCBTI) (Experimental): Based on the existing consensus concerning non-pharmacological treatment of insomnia, Hvil® includes the following treatment components: sleep hygiene, sleep optimization, stimulus control therapy, deactivation/relaxation training, and cognitive therapy. Intervention duration is approximately six to nine weeks.
  Interventions: Behavioral: Digitally delivered CBTI (eCBTI)

INTERVENTIONS:
Behavioral: Digitally delivered CBTI (eCBTI) — Based on the existing consensus concerning non-pharmacological treatment of insomnia, Hvil® includes the following treatment components: sleep hygiene, sleep optimization, stimulus control therapy, deactivation/relaxation training, and cognitive therapy. Intervention duration is approximately six to nine weeks.
  Arms: Digitally delivered CBTI (eCBTI)

SUMMARY:
Insomnia is a widespread public health challenge considering its impact on daily life, comorbidity with other disorders, and socio-economic costs. Previous research has shown the efficacy of cognitive behavioral therapy for insomnia (CBTI), and recent research indicates that digitally delivered CBTI (eCBTI) is highly efficacious, and statistically significantly equivalent to in-person delivered CBTI (ipCBTI) for treating insomnia. However, research is limited as to how eCBTI can be integrated into general practice as a non-pharmacological alternative to hypnotics. This study aims to evaluate the feasibility, acceptability, and effectiveness of a fully automated mobile application for treating insomnia in general practice. The secondary aims are to examine effects on psychological and physical comorbidities, possible moderators and mediators of the effect of eCBTI, and cost-effectiveness.

DETAILED DESCRIPTION:
Insomnia is prevalent in the general population (10%) and particularly so among patients in general practice (30-50%), with considerable costs to the individual and society. Hypnotics, which remain the most common treatment option in general practice, are usually not curative and are associated with risks of side effects, dependence, tolerance, and increased mortality. In contrast, cognitive behavioral therapy for insomnia (CBTI) has been shown to be highly efficacious and is recommended as the first-line treatment for insomnia by organizations such as the American Academy of Sleep Medicine, the American College of Physicians, and the European Sleep Research Society.

However, the challenge remains to make CBTI available to meet population needs due to several barriers, including a limited number of trained therapists, the costs of delivering CBTI face-to-face, and physical and geographical constraints. Digitally delivered CBTI (eCBTI) has been shown to be a possible approach to overcoming these challenges, but research on the effectiveness of eCBTI in a general practice setting remains limited.

Given the current lack of non-pharmacological treatment options for insomnia in general practice and the considerable potential of eCBTI to treat insomnia, the primary aim of the proposed study is to evaluate the feasibility, acceptability, and short- and longer-term efficacy of eCBTI for the treatment of insomnia in general practice. Our secondary aims are: a) to evaluate the possible benefits of treating insomnia on psychological and physical symptoms and comorbidities, b) to explore for whom the intervention works by examining the possible moderating effects of information technology proficiency and socio-demographic, clinical, and work-related factors, c) to investigate the possible working mechanisms, including changes in sleep-related cognitions and behaviors, and d) to assess the cost-effectiveness of the intervention.

The study is designed as a cluster-randomized controlled trial, randomizing general practitioners (GPs) from three Danish regions to screen patients for insomnia and offer either hvil®, a mobile-based program for delivering CBTI (eCBTI), or care as usual to those with moderate to-severe insomnia (ISI ≥ 10). A total of 2 X 50 GPs are expected to recruit a minimum of 2 X 250 patients who will complete the intervention. The intervention lasts 10 weeks, including an initial one-week assessment period.

The primary outcome is insomnia severity, assessed with the Insomnia Severity Index (ISI). Secondary sleep diary-based outcomes include sleep onset latency (SOL), wake after sleep onset (WASO), total sleep time (TST), time in bed (TiB), and sleep efficiency (SE). Secondary non-sleep outcomes include quality-of-life (QoL) and psychological and physical symptoms such as anxiety, depression, fatigue, and pain. Cost-effectiveness will be assessed using data on healthcare utilization, social benefits, and employment from Danish national registries. Outcomes will be assessed at baseline (week 0) (T1), halfway through the intervention (week 5), post-intervention (week 11) (T3), and follow-up (6 months) (T4).

Baseline group differences (concerning socio-demographic, disease-related, and psychosocial data) will be explored to test the success of the randomization. If differences are found, sensitivity analyses will be made to evaluate their possible influence on the results. Main effects will be analysed using Mixed Linear Models (MLMs) based on the intent-to-treat sample. MLMs account for the hierarchical, non-independent nature of the data (i.e., repeated measures nested within patients and treatment conditions), testing the time*group interaction effect, reflecting the effect of treatment. Moderation analyses will evaluate whether individual differences in various baseline variables (e.g., physical function, expectations, computer proficiency, chronotype, etc.) or treatment adherence influence intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Individuals who report moderate-to-severe insomnia symptoms (a score ≥10 on the Insomnia Severity Index, ISI)
* Individuals referred by their general practitioner
* Individuals with access to a smartphone with internet connection
* Individuals who report sufficient technological proficiency (e.g., ability to download apps)

Exclusion Criteria:

* Children (<18 years)
* Individuals who report mild or no clinically relevant insomnia symptoms (a score <10 on the ISI)
* Individuals who have a shift-work schedule or are on maternity/paternity leave
* Individuals who are unable to read Danish
* Individuals who report severe physical or psychological comorbidity with known effects on sleep (e.g., psychosis, cancer, COPD)
* Individuals who report other diagnosed sleep or circadian rhythm disorders (e.g., sleep apnea, narcolepsy)
* Individuals who are currently receiving or have recently received CBTI or eCBTI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the Insomnia Severity Index (ISI), with scores ranging from 0 to 28, where higher scores indicate higher insomnia severity, and a score equal to or above 10 indicates clinical significance.

SECONDARY OUTCOMES:
Sleep diary outcomes | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the Consensus Sleep Diary (CSD), which measures sleep- and waking time, sleep onset latency (SOL), wakefulness after initial sleep onset (WASO), early morning awakenings (EMA), and risetime, allowing for total sleep time (TST), total time in bed (TIB), and sleep efficiency (SE) to be calculated.
Sleep quality | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the Pittsburgh sleep quality index (PSQI), which measures clinically derived domains of sleep difficulties (i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction).
Daytime fatigue | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the Functional Assessment of Chronic Illness Therapy for Fatigue (FACIT-Fatigue), which covers physical fatigue, functional fatigue, and social consequences of fatigue.
Cognitions about sleep | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16).
Physical and mental functioning | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the Short Form Health Survey (SF-12), which addresses different aspects of emotional states and daily activities. The questionnaire allows for sub-scores for mental and physical health to be calculated based on population norms, with higher scores indicating better health
Psychological distress | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the Depression, Anxiety, and Stress Scales-21 (DASS-21), which evaluates the constructs depression, anxiety, and stress on sub-scales.
Health-related well-being | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the 5-item World Health Organisation&amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s Well-Being Index (WHO-5).
Application usability | Post-treatment (approximately week 11)
  Assessed with the short version of the mHealth App Usability Questionnaire (MAUQ-S).
Health-related quality of life | Baseline (week 0), post-treatment (approximately week 11), follow-up (approximately week 37)
  Assessed with the five-dimensional EuroQol (EQ-5D-5L), which measures self-reported health and well-being across five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, as well as overall health on a 0-100 VAS. A higher score indicates better quality of life.
Socio-economic costs | Throughout the study period, from study enrollment (week 0) to follow-up at 37 weeks
  Assessed with data from Danish national registers on redeemed medicine prescriptions, use of primary and secondary health care services, long-term sickness absence

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, Professsor, DMSc, MSc, Principal Investigator — University of Aarhus and Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the study will be made available in an irreversibly anonymized form. However, only data of those participants can be shared who have explicitly given consent to this as part of their informed consent to study participation. This means that it may not be possible to share all data underlying a certain publication. Data will be shared exclusively for research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No later than six months after publication, no end date.
Access Criteria: Data will be shared exclusively with other researchers and for research purposes only. Researchers requesting the data will have to provide a methodologically sound research proposal clarifying how the data will be used and for what purpose.